CLINICAL TRIAL: NCT03215511
Title: A Phase 1 Study of the TRK Inhibitor Selitrectinib (BAY 2731954) in Adult and Pediatric Subjects With Previously Treated NTRK Fusion Cancers
Brief Title: A Study to Test the Safety of the Investigational Drug Selitrectinib in Children and Adults That May Treat Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20810; LOXO-EXT-17005 (Other: Loxo Oncology, Inc.); 2017-004246-20 (EudraCT Number)
Expanded Access: NCT03206931 (No longer available)
Record Dates: First submitted 2017-06-30; First posted 2017-07-12 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Solid Tumors Harboring NTRK Fusion
Keywords: Solid Tumor; Metastatic cancer; Advanced cancer; Neurotrophic tyrosine receptor kinase (NTRK); NTRK1; NTRK2; NTRK3; Fusion Positive; Children
MeSH Terms: conditions — Neoplasm Metastasis | interventions — selitrectinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cancer participants <12 years (Experimental): A Rolling-6 dose escalation design will be used. The starting dose for participants age < 12 years will be 25% below the highest dose level cohort divided by 1.73 m^2 cleared by the Safety Review Committee (SRC) for subjects age 12 years and older.
  Interventions: Drug: Selitrectinib (BAY2731954)
- Cancer participants ≥12 years (Experimental): A 3+3 dose escalation design will be used to determine the maximum tolerated dose (MTD)/recommended dose for further study, enrolling 3 to 6 participants per cohort with a starting dose level of 100 mg twice daily (BID).
  Interventions: Drug: Selitrectinib (BAY2731954)

INTERVENTIONS:
Drug: Selitrectinib (BAY2731954) — Selitrectinib is administered as capsules or liquid formulation.
  Other Names: Loxo-195

SUMMARY:
This research study is done to test the safety of the new drug selitrectinib in children and adults with cancer having a change in a particular gene (NTRK1, NTRK2 or NTRK3). The drug may treat cancer by interfering with the effect of the NTRK genes on cancer growth. The study also investigates how the drug is absorbed and processed in the human body, and how well and for how long the cancer responds to the drug. This is the first study to test selitrectinib in humans with cancer, for whom no other effective therapy exists.

DETAILED DESCRIPTION:
The primary objective is to determine the recommended dose for further study of oral selitrectinib with previously treated neurotrophic tyrosine kinase (NTRK) cancers in 2 patient groups: a) aged 12 years and older and b) younger than 12 years. Secondary objectives of Phase I are to characterize the pharmakokinetic properties of the test drug, its safety and tolerability, and to assess the objective response rate (ORR) of NTRK-tumors.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumor for which, in the opinion of the investigator, no other standard therapy offers greater benefit.
* A solid tumor diagnosis in the setting of:

  * a) a documented NTRK fusion and a clinical history of relapse following a response to a prior TRK inhibitor
  * b) a documented NTRK fusion unresponsive to a prior TRK inhibitor
  * c) a documented NTRK fusion and a clinical history of intolerance to a prior TRK inhibitor
* NTRK gene fusions will be identified in a CLIA-certified (or equivalently-accredited diagnostic) laboratory. If such a report cannot be provided, other available certifications/accreditations are required and need to be documented. Patients with infantile fibrosarcoma (IFS) or congenital mesoblastic nephroma (CMN) may be enrolled based on an ETV6+ FISH test without identifying NTRK3.
* Performance Status: Eastern Cooperative Oncology Group (ECOG) score ≤ 2 in adults or Karnofsky Performance Status (KPS) Score≥50% (age ≥ 16 years) or Lansky Performance Score (LPS) ≥ 40% (age < 16 years).
* Life expectancy of at least 3 months.
* Adequate hematologic, hepatic and renal function.
* Patients with stable central nervous system (CNS) primary tumor, brain metastases, or treated spinal cord compression are eligible if neurological symptoms have been stable for 7 days prior to the first dose of selitrectinib.
* Ability to receive study drug orally or by enteral administration

Exclusion Criteria:

* Prior exposure to second generation TRK inhibitor (e.g. selitrectinib, repotrectinib [TPX-0005]), taletrectinib [DS-6501b/AB-106]). Exception is in case patient presented intolerance to the second generation TRK inhibitor agent and the duration of exposure was less than 28 days. No previous treatment with selitrectinib is allowed.
* Concurrent treatment with a strong CYP3A4 inhibitor or inducer, consumption of grapefruit juice or Seville oranges, or drugs associated with QT prolongation.
* Clinically significant active cardiovascular disease or history of myocardial infarction within 3 months prior to planned start of selitrectinib, or prolongation of QT interval corrected for heart rate (QTc interval) >480 milliseconds within past 6 months
* Major surgery within 7 days of enrollment
* Uncontrolled systemic bacterial, fungal or viral infection.
* Pregnancy or lactation.
* Known hypersensitivity to selitrectinib or Ora-Sweet® SF and OraPlus® for patients receiving liquid formulation.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Up to 42 days
Recommended dose | Up to 12 months

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 56 months
Severity of adverse events | Up to 56 months
  Severity is assessed using CTCAE version 4.03
Duration of adverse events | Up to 56 months
Number of subjects with safety-relevant changes in clinical parameters or vital signs after drug administration | Up to 56 months
Severity of safety-relevant changes in clinical parameters or vital signs after drug administration | Up to 56 months
Overall response rate (ORR) in subjects with NTRK fusion cancer previously treated with TRK inhibitor determined by investigator | Up to 56 months
  ORR is determined by the investigator using the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Overall response rate (ORR) in subjects with primary central nervous system (CNS) malignancies determined by investigator | Up to 56 months
  ORR is determined by the treating investigator using the Response Assessment in Neuro-Oncology (RANO) criteria.
Maximum concentration (Cmax) of BAY2731954 in plasma | Predose, 0.25, 0.5, 1, 2, 4, 6, 8 hours post-dose on Day 1, predose, 0.5, 1, 2, 4 post-dose on Day 8 of Cycle 1 (cycle length 28 days)
Area under the concentration versus time curve of BAY2731954 in plasma (AUC (0-10), AUC(0-12) for BID dosing and AUC(0-24) for QD dosing) | At defined time points for different cohort, up to 10 hours post-dose

CONTACTS AND LOCATIONS:
Locations (29):
- United States (17):
  - Univ.of California-San Diego Moores Cancer Center, La Jolla, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Stanford Cancer Center, Palo Alto, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Midwestern Regional Medical Center, Zion, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Sydney Children's Hospital, Sydney, New South Wales
  - Royal Children's Hospital Melbourne, Parkville, Victoria
- UZ Antwerpen, Edegem, Belgium
- Rigshospitalet - Kræftbehandling, Copenhagen, Denmark
- France (2):
  - Institut Curie - Ulm - Paris, Paris
  - Institut Gustave Roussy - Département de Médecine Oncologique, Villejuif
- Universitätsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg, Germany
- Tallaght Hospital, Dublin, Ireland
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy, Italy
- National Cancer Center Singapore, Singapore, Singapore
- Spain (2):
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Fundacion Jimenez Diaz (Clinica de la Concepcion), Madrid

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] O'Reilly EM, Hechtman JF. Tumour response to TRK inhibition in a patient with pancreatic adenocarcinoma harbouring an NTRK gene fusion. Ann Oncol. 2019 Nov 1;30(Suppl_8):viii36-viii40. doi: 10.1093/annonc/mdz385. Epub 2019 Dec 24. PMID 31605106
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards — https://clinicaltrials.bayer.com/study/20810
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/